CLINICAL TRIAL: NCT01484392
Title: Determinants of Compliance With Glaucoma Therapy
Status: Completed | Type: Observational
Sponsor: Legacy Health System (Other)
Responsible Party: Principal Investigator, Steven L. Mansberger, Associate Scientist, Legacy Health System
Other Study IDs: FWA00001280
Record Dates: First submitted 2011-11-30; First posted 2011-12-02 (Estimated); Last update posted 2016-03-09 (Estimated); Status verified 2016-03

CONDITIONS: Open Angle Glaucoma
Keywords: open angle glaucoma; compliance; adherence
MeSH Terms: conditions — Glaucoma, Open-Angle; Patient Compliance

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to determine which medical, demographic, and health belief factors are associated with glaucoma therapy compliance.

ELIGIBILITY:
Inclusion Criteria:

* open angle glaucoma
* be well controlled on current medical therapy
* be using a prostaglandin analogue

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with open angle glaucoma.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2006-08; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Compliance with glaucoma medication at 1 month | 1 month after enrollment
  Compliance is measured using the Travatan Dosing Aid, a device that records when patients administer their topical glaucoma medication.
Compliance with glaucoma medication at 3 months | 3 months after enrollment
  Compliance is measured using the Travatan Dosing Aid, a device that records when patients administer their topical glaucoma medication.

CONTACTS AND LOCATIONS:
Overall Officials: Steven L Mansberger, MD, MPH, Principal Investigator — Legacy Health
Locations (1):
- Devers Eye Institute, Portland, Oregon, United States